CLINICAL TRIAL: NCT01627769
Title: Comparison of the Blister Fluid Components of Second Degree Burned Patients With the Blister Fluid Components Following Intralesional Cryosurgery of Keloid Scars - A Feasibility Study.
Brief Title: Evaluation and Comparison of Keloids and Second Degree Burns Blisters Fluid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Yaron Har-Shai, Professor, Carmel Medical Center
Other Study IDs: CMC-12-0050-CTIL
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Blisters; Second Degree Burns; Wounds
Keywords: scars; blisters; second degree burns; cryosurgery; keloid scars; hypertrophic scars
MeSH Terms: conditions — Blister; Wounds and Injuries; Cicatrix; Keloid; Cicatrix, Hypertrophic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blister fluid of kryosurgery and second degree burns Following the results of the above study a further extension of the study is progressing in which the identification of the cell population in the blister fluid following intralesional cryosurgery of keloid scars is examined
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- second degree blisters patients: blister fluids of second degree burns
- cryotherapy blisters: blister fluids of cryosurgery wounds

SUMMARY:
It is well documented that following thermal burns injury the development of hypertrophic scars and keloid (HSK) ranges between 40 to 90%. on the other hand It is well documented that cryosurgery wounds generally heal with minimal tissue contraction, resulting in good cosmetic results and with minimal complications.

The Aim of the study is To specify the burn and cryosurgery blister fluid for proteins, cytokines and cells and To compare between the above data regarding possible proteins, cytokines and cells, in regard to their possible effect on scarring and wound healing.

Also to Identify those components which are present only in the cryosurgery blister and which might have an anti-scarring effect and to characterize them biochemically.

DETAILED DESCRIPTION:
Skin is the most frequently injured tissue, and millions of people worldwide acquire scars every year. Clinical experience shows that patients want less noticeable scars, with color and texture that closely resemble their normal skin.

Few humans reach adulthood without experiencing a wound to the skin that result in a scar. Scars range from fine lines to raised, hard, red, pruritic and painful hypertrophic or keloid scars, which are severely disfiguring and cause significant morbidity. In addition to physical complications, the appearance of scars can be a major concern for both physicians and their patients. Published literature shows that wide demographic groups, across gender, age, ethnicity and geographical region, have similar concerns about scarring and that patients, in particular, value even small improvements in scarring. It is well established that severe and disfiguring scarring can be associated with significant psychological stress and impairment of quality of life .

It is well documented that following thermal burns injury the development of hypertrophic scars and keloid (HSK) ranges between 40 to 90%.

In the second degree burn the exudate accumulates locally between the epidermis and the dermis of skin, forming blisters. Burn exudate (blister) forms as a result of changed capillary permeability when the damaging agent locally affects the capillaries, as it generally does in inflammatory reactions.

The chemical composition of exudate is very like that of plasma, the protein concentration depending on the degree of damage in capillaries. Further, exudate contains material from damaged and disintegrated cells such as protein degradation products, enzymes etc. By puncturing blisters it should be possible to follow the changes in their content during the healing process.

Only few studies were published in the medical literature in which the blister fluid composition was evaluated following a second degree burn. Nanto and Viljanto at 1962 were the first to publish the chemical composition of blister fluid. They have demonstrated that the albumin-globulin ratio, the phosphorus content and the quantity of purines and pyrimidine derivatives in the blister fluid can be indicators of the local severity of second degree burn.

Heggers et al in 1980 have found that blister fluid, following burn, contained all substances found in the body, including parenterally administered penicillin. In addition the elevation of potassium and the cation to anion imbalance is primarily due to the Na/K cellular pump malfunction, and the destruction of the permeability of the cell membrane is most likely a direct result of complement and other cellular enzymes, which include prostaglandins and thromboxane. Elevated SGOT, CPK, and LDH enzymes indicate severe trauma to the cells. The presence of immunoglobulins indicate that high molecular-weight proteins diffuse equally well during this edematous phase.

In 1986 Deitch et al. studied early protein alteration in the blister fluid and serum associated with burn injury. It was found that local changes in the blister fluid may adversely affect local immunity and predispose the patient to burn wound sepsis.

Lately, a significant improvement in protein identification employing proteomic profiling technology has been documented. The model which is used is the suction blister fluid which is compared with protein expression in pathological skin conditions such as psoriasis and toxic epidermal necrolysis.

However, the evaluation of the blister fluid components on cutaneous scarring has not been investigated.

In 1982, Shepherd and Dawber were the first to apply cryosurgery as a monotherapy regimen for treating Hypertrophic scars and keloids (HSK). Mende, Zouboulis and Orfanos and others showed that repeated surface/spray cryosurgical sessions can have a beneficial effect on HSK (between 68% - 81% remission), with almost no recurrence (2%).

Recently, an intralesional cryosurgery technology has been developed to treat HSK (CryoShape, Etgar Group International Ltd., Kefar Saba, Israel approved by the Israel ministry of Health) (14-21). A specially designed cryoneedle is inserted into the core of the HSK so as to maximize the volume of the HSK to be frozen. The cryoneedle is connected by an adaptor to a cryogun filled with liquid nitrogen, which is introduced into the cryoprobe thereby freezing the HSK. After the HSK is completely frozen, the cryoprobe defrosts and is withdrawn.

Following the cryotreatment a blister is formed. It has been demonstrated that an average of 51 % of scar volume reduction was achieved following a single intralesional cryosurgery treatment. Specifically, for auricular and lobular HSK the average volume reduction was 67% and for upper back and shoulders HSK 60%. These obtained clinical results are significant superior to any other treatment modalities which exist now-days to treat HSK.

Scientific studies which have been executed following the intralesional cryosurgery treatment have demonstrated rejuvenation of the treated scars, i.e., parallelization, and a more organized architecture of the collagen fibers when compared to the pre-treated scars. In addition, histological analysis revealed that after intralesional cryosurgery the collagen bundles lost their swirl structure, the thickness of the collagen layer decreased, and the bundles became more compact with less space between the fibers. A clear distinct transition zone separated the treated from the unaffected area. The frozen tissue was devoid of proliferating cells and of mast cells whereas the number of blood vessels remained unaltered. Most of the fibroblasts expressed all tested myofibroblast markers although some of them exclusively expressed one and not the other. Almost no mast cells were found following the cryo-treatment. Thus, Intralesional cryosurgery treatment resulted in major changes in collagen structure and organization. In addition, the treatment reduced the numbers of proliferated cells in general and myofibroblasts and of mast cells in particular.

It is well documented that cryosurgery wounds generally heal with minimal tissue contraction, resulting in good cosmetic results and with minimal complications.

However, following an extensive medical literature search it has been evident that the evaluation of the blister fluid components following skin cryosurgery for the treatment of HSK has not yet been studied as well as the specific evaluation of post-cryosurgery blister components on cutaneous scarring/anti-scarring effect.

ELIGIBILITY:
Inclusion Criteria:

1. subject agrees to enroll in the research
2. subject provides written authorization for use and disclosure of protected health information
3. subject provides written informed consent
4. subject who suffer a second degree burn with intact blisters from hot water or liquid within 24 hours, and have been admitted to the emergency room at Carmel Medical center
5. subject suffering from keloids and are treated at the Department of Plastic Surgery , Linn Medical Center, by the intralesional cryosurgery method within the last 24 hours and have developed an intact blister

Exclusion Criteria:

1. subject who has a blister exudate that is culture positive
2. subject who has any signs of infection in and/or around the blister
3. subject with blisters present more then 24 hours (after which samples will not be taken)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with second degree burns patients status post cryosurgery treatment for keloid scars with post treatment blisters
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-07; Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
comparison of inflamation cells and proteins (proteomic evaluation) between blisters caused by heat and blisters caused by cryo injury | at time of sampling.
  the protein evaluation and comparison is achieved by the use of proteomic study which evaluate the quantity of about 700 different proteins in the fluid of the different blisters (heat blisters compared to "cryo" blisters).
  we also evaluate the differences in quntities between the inflamation cells in each sample.

CONTACTS AND LOCATIONS:
Overall Officials: yaron har-shai, Md, Principal Investigator — carmel medical center- ISRAEL
Locations (1):
- Carmel Medical Center, Haifa, Haifa District, Israel